CLINICAL TRIAL: NCT01400139
Title: An Open-label, Multicenter Study to Assess the Long -Term Safety of Hydrocodone Bitartrate (HYD) Tablets 20 to 120 mg Once-daily in Subjects With Moderate to Severe Chronic Nonmalignant and Nonneuropathic Pain
Brief Title: Long-term Safety of Once-daily Hydrocodone Bitartrate (HYD) Tablets For Moderate to Severe Chronic Nonmalignant and Nonneuropathic Pain. Includes a 24-week Extension Period.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYD3003
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Nonmalignant and Nonneuropathic Pain
Keywords: Pain; Nonmalignant pain; Nonneuropathic Pain; Opioid
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydrocodone bitartrate (Experimental): Hydrocodone bitartrate (HYD) once daily (q24h) tablets
  Interventions: Drug: Hydrocodone bitartrate q24h film-coated tablets

INTERVENTIONS:
Drug: Hydrocodone bitartrate q24h film-coated tablets — Hydrocodone bitartrate q24h film-coated tablets 20 - 120 mg once daily
  Other Names: Hysingla ER

SUMMARY:
The primary objective of this study is to characterize the long-term safety of Hydrocodone Bitartrate (HYD) tablets 20 to 120 mg once-daily in subjects with chronic nonmalignant and nonneuropathic pain.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects ≥ 18 years of age with moderate to severe, chronic nonmalignant and nonneuropathic pain (lasting several hours daily) as their predominant pain condition for at least 3 months prior to the screening visit;
* Subjects deemed by the investigator/medically qualified designee (must be MD or DO) to be appropriate candidates for the protocol specified, around the clock HYD therapeutic regimen;
* Female subjects who are premenopausal or postmenopausal less than 1 year and who have not had surgical sterilization (ie, tubal ligation, partial or complete hysterectomy) must have a negative serum pregnancy test, be nonlactating, and willing to use adequate and reliable contraception throughout the study (eg, barrier with additional spermicidal foam or jelly, intra-uterine device, hormonal contraception);
* Subjects who are willing and able to be compliant with the protocol, are capable of subjective evaluation (ie pain scores), are able to read and understand questionnaires, are willing and able to use an electronic diary, and are able to read, understand, and sign the written informed consent form in English.

Exclusion Criteria include:

* Subjects taking opioid analgesic(s) equivalent to > 120 mg/day of oxycodone during the 14 days prior to the screening visit;
* Subjects who previously participated in an investigational hydrocodone study within 90 days prior to the first dose of study medication ;
* Subjects who have used any investigational medication other than hydrocodone within 30 days prior to the first dose of study drug;
* Subjects with any history of seizures (subjects with history of pediatric febrile seizures may participate in the study) or increase in intracranial pressure;
* Subjects with current uncontrolled depression or other uncontrolled psychiatric disorder (subjects with controlled depression or other psychiatric disorder must be on a stable medication for ≥ 1 month prior to the screening visit to participate in the study);
* Subjects with a history of alcohol, medication, or illicit drug abuse or addiction and/or history of opioid abuse or addiction at any time;
* Subjects with clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling pacemaker;
* Subjects with unstable respiratory disease that, in the opinion of the investigator, precludes entry into this study;
* Subjects with biliary tract disease, hypothyroidism, adrenal cortical insufficiency, or any other medical condition that, in the opinion of the investigator, is inadequately treated and precludes entry into the study;
* Subjects with history of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated;
* Subjects with evidence of impaired liver function upon entry into the study (laboratory test values ≥ 3 times the upper limit of the laboratory reference (normal) range (ULN) for aspartate transaminase [AST/SGOT] or alanine transaminase [ALT/SGPT], or values > 2 times the ULN for alkaline phosphatase), or total bilirubin level > 1.5 times the ULN or, in the opinion of the investigator/medically qualified designee (must be MD or DO), liver function impairment to the extent that the subject should not participate in this study;
* Subjects with evidence of impaired kidney function upon entry into the study (ie, serum creatinine ≥ 2.5 mg/dL);
* Subjects with any condition in which opioids are contraindicated, eg, severe respiratory depression with hypoxia and/or hypercapnia, severe chronic obstructive lung disease, cor pulmonale, severe bronchial asthma, or paralytic ileus;
* Subjects who are allergic to hydrocodone or who have a history of allergies to other opioids. This does not include subjects who have experienced common opioid side effects (eg, nausea, constipation);
* Subjects receiving monoamine oxidase inhibitors (MAOIs) or who have been taking MAOIs within 2 weeks of the screening visit.

Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (98):
  - Alliance Clinical Research, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - ACRI -Phase1, LLC, Anaheim, California
  - United Clinical Research Center, Inc., Anaheim, California
  - Med Center, Carmichael, California
  - Research Center of Fresno, Inc., Fresno, California
  - TriWest Research Associates, La Mesa, California
  - Torrance Clinical Research, Lomita, California
  - Skyline Research, LLC, Long Beach, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Center for Clinical Research, Inc, Richmond, California
  - Northern California Research, Sacramento, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Meridien Research, Bradenton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Neuroscience Consultants LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - Atlanta Knee and Shoulder Clinic, PC, Stockbridge, Georgia
  - Illinois Center for Clinical Research, Chicago, Illinois
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - ICRI, Leawood, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Advance Clinical Research, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Research Facility, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - CRI Worldwide LLC, Willingboro, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Research Across America, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Daystar Clinical Research, Inc., Akron, Ohio
  - IVA Research, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Bone Joint and Spine Surgeons, Inc., Toledo, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Allegheny Pain Management, P.C., Altoona, Pennsylvania
  - Pennsylvania Research Institute, Bensalem, Pennsylvania
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Tipton Medical & Diagnostic Center, Tipton, Pennsylvania
  - Hartwell Research Group, Anderson, South Carolina
  - Pain Research of Charleston, Charleston, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Heartland Medical, PC, New Tazewell, Tennessee
  - HCCA Clinical Research Solutions, Smyrna, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Lovelace Scientific Resources, Inc., Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - Heights Doctor's Clinic, Houston, Texas
  - JVC Family Medicine, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - TEAM Research of Central Texas, Killeen, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Sun Research Institute, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Aspen Clinical Research, Orem, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - HypotheTest, LLC, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Washington Center for Pain Management, Edmonds, Washington

REFERENCES:
- [Result] Wen W, Taber L, Lynch SY, He E, Ripa S. 12-Month safety and effectiveness of once-daily hydrocodone tablets formulated with abuse-deterrent properties in patients with moderate to severe chronic pain. J Opioid Manag. 2015 Jul-Aug;11(4):339-56. doi: 10.5055/jom.2015.0283. PMID 26312961
- [Derived] Campbell K, Kutz JW Jr, Shoup A, Wen W, Lynch SY, He E, Ripa SR. Evaluation of the Ototoxicity Potential of Once-Daily, Single-Entity Hydrocodone in Patients with Chronic Pain: Results of Two Phase-3 Clinical Studies. Pain Physician. 2017 Jan-Feb;20(1):E183-E193. PMID 28072811
- [Derived] Kapil RP, Cipriano A, Wen W, Yu Lynch S, He E, Colucci SV, Harris SC. Pharmacokinetic Profile and Sustained 24-hour Analgesia of a Once-daily Hydrocodone Bitartrate Extended-release Tablet with Abuse-deterrent Properties. Clin Ther. 2016 Feb;38(2):302-14. doi: 10.1016/j.clinthera.2015.12.003. Epub 2015 Dec 31. PMID 26749219
- [Derived] Taber L, Lynch SY, He E, Ripa SR. Long-term safety and effectiveness of once-daily, single-entity, extended-release hydrocodone over 76 weeks of an open-label study in patients with chronic noncancer and nonneuropathic pain. Postgrad Med. 2016 Jan;128(1):23-33. doi: 10.1080/00325481.2016.1134022. Epub 2016 Jan 12. PMID 26681111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Core study: First subject first visit: 22-July-2011; Last subject last visit: 26-August-2013. Extension period: First subject first visit: 24-April-2013; Last subject last visit of 24-February-2014. The Core and Extension studies were conducted at medical/research sites in the United States.
Pre-assignment Details: Subjects with moderate to severe, chronic nonmalignant and non-neuropathic pain.
Groups:
- Hydrocodone Bitartrate (HYD): Hydrocodone bitartrate (HYD) once daily (q24h) tablets
  Hydrocodone bitartrate q24h film-coated tablets: Hydrocodone bitartrate q24h film-coated tablets 20 - 120 mg once daily
Period: HYD Core Study
Arm/Group | Hydrocodone Bitartrate (HYD)
Started | 922
Completed | 410
Not Completed | 512
Not completed — Adverse Event | 210
Not completed — Lack of Efficacy | 59
Not completed — Withdrawal by Subject | 114
Not completed — Lost to Follow-up | 39
Not completed — Confirmed or suspected diversion | 20
Not completed — Administrative | 56
Not completed — Did not qualify for Maintenance Period | 14
Period: HYD Extension Period
Arm/Group | Hydrocodone Bitartrate (HYD)
Started | 106 (Subjects completing the Core Study were offered an option to enter the 24-week open-label Extension)
Completed | 83
Not Completed | 23
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 5
Not completed — Administrative | 10

BASELINE CHARACTERISTICS:
Groups:
- HYD Core Study: Hydrocodone bitartrate (HYD) once daily (q24h) tablets
  Hydrocodone bitartrate q24h film-coated tablets: Hydrocodone bitartrate q24h film-coated tablets 20 - 120 mg once daily
Arm/Group | HYD Core Study
Number analyzed (Participants) | 922
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 526
  Male | 396
Race/Ethnicity, Customized [Number; unit: participants]
  White | 761
  Black or African American | 141
  Native Hawaiian or other Pacific Islander | 2
  Asian | 8
  American Indian or Alaska Native | 4
  Other | 6
Screening Baseline Pain Over the Last 24 Hours [Mean (Standard Deviation); unit: units on a scale] — "Average pain over the last 24 hours" score (on an 11-point numerical rating scale where 0 = no pain and 10 = pain as bad as you can imagine).
  units on a scale | 6.4 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety
Description: Safety assessments included AEs, clinical laboratory test results, vital sign measurements, ECG findings, and audiology assessments.
Time Frame: Up to 84 weeks
Population: The Core Study safety population (N=922) was defined as the group of subjects who received at least 1 dose of study drug during the study. The Extension Period safety population (N=106) was the group of core study safety population subjects who entered the extension period and received at least 1 dose of study drug in the extension period.
Measure: Number; unit: participants
Groups:
- HYD Extension Period: Hydrocodone bitartrate (HYD) once daily (q24h) tablets
  Hydrocodone bitartrate q24h film-coated tablets: Hydrocodone bitartrate q24h film-coated tablets 20 - 120 mg once daily
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 922 | 106
participants
  Serious adverse events | 80 | 6
  All other adverse events in ≥ 5% of patients | 586 | 0

2. Primary Outcome: Daily "Average Pain Over the Last 24 Hours"
Description: "Average pain over the last 24 hours" score (on an 11-point numerical rating scale where 0 = no pain and 10 = pain as bad as you can imagine).
Time Frame: Core study: from start to end of maintenance period (up to 52 weeks); Extension study: from start of maintenance to end of extension (up to 76 weeks)
Population: The Core Study population analyzed (N=727) was the group of subjects who received at least 1 dose of study drug during the maintenance period. The Extension Period population analyzed (N=106) was the group of core study safety population subjects who entered the extension period and received at least 1 dose of study drug in the extension period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 727 | 106
units on a scale | 3.6 (1.80) | 3.8 (1.73)

3. Secondary Outcome: "Pain Right Now" Score
Description: "Pain right now" scores were collected using an 11-point scale where 0 = no pain and 10 = pain as bad as you can imagine. The "pain right now" scores were only collected during the Core Study. "Pain right now" scores were not assessed during the Extension Period.
Time Frame: Week 12
Population: The Core Study population analyzed was the group of subjects who received at least 1 dose of study drug during the maintenance period and provided data. Data were not collected for this outcome measure during the Extension Period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 723 | 0
units on a scale | 3.46 (0.071) |

4. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Scale - Revised (MOS Sleep-R)
Description: The MOS Sleep-R is a brief, self-administered 12-item assessment designed to measure key aspects of sleep. It includes a sleep problems index II and 6 subscale scores - sleep disturbance, sleep adequacy, daytime somnolence, snoring, awaken short of breath or with headache, and quantity of sleep. For each individual and time of assessment, quantity of sleep was recorded as the number of hours slept per night. The number of hours it took the subject to fall asleep per night was categorized 1, 2, 3, 4, or 5 corresponding to 0 through 15, 16 through 30, 31 through 45, 46 through 60, or more than 60 minutes, respectively. The other scales were recorded as 1 = all of the time, 2 = most of the time, 3 = some of the time, 4 = a little of the time, or 5 = none of the time. A higher value indicates a better score, therefore a positive change from baseline indicates a better sleep pattern and a negative change from baseline indicates a worsening in sleep pattern.
Time Frame: Baseline and up to 52 weeks in the Core Study maintenance period, and up to 24 weeks in the Extension Period
Population: The Core Study population analyzed was the group of subjects who received at least 1 dose of study drug during the maintenance period and provided data. The Extension Period safety population was the group of core study safety population subjects who entered the extension and received at least 1 dose of study drug in the extension period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 718 | 106
units on a scale
  Change from Baseline in Sleep Disturbance: number analyzed (Participants) | 710 | 106
  Change from Baseline in Sleep Disturbance | 4.69 (8.276) | 3.65 (7.993)
  Change from Baseline in Sleep Adequacy: number analyzed (Participants) | 710 | 106
  Change from Baseline in Sleep Adequacy | 3.29 (8.959) | 2.94 (8.264)
  Change from Baseline in Daytime Somnolence: number analyzed (Participants) | 710 | 106
  Change from Baseline in Daytime Somnolence | 0.57 (8.469) | 0.89 (8.418)
  Change from Baseline in Snoring: number analyzed (Participants) | 710 | 106
  Change from Baseline in Snoring | 1.28 (6.839) | 1.77 (6.960)
  Change from Baseline in Shortness of Breath: number analyzed (Participants) | 710 | 106
  Change from Baseline in Shortness of Breath | 1.46 (9.788) | 3.46 (10.109)
  Change from Baseline in Quantity of Sleep: number analyzed (Participants) | 710 | 106
  Change from Baseline in Quantity of Sleep | 0.29 (1.413) | 0.17 (1.189)
  Change from Baseline in Sleep Problem Index II: number analyzed (Participants) | 710 | 106
  Change from Baseline in Sleep Problem Index II | 4.04 (8.530) | 3.70 (8.248)

5. Secondary Outcome: Brief Pain Inventory Short Form (BPI-SF)
Description: The BPI-SF assessed the severity of pain and interference of pain on daily functions. It consists of 9 sections denoted by Q1 to Q8 and Q9A to Q9G according to their order in the questionnaire, that measure pain location, intensity, pain treatment, and functional interference of pain on mood and every day activities. Scores ranged from 0 (none) to 10 (worst as can be). Four of the items (questions 3 to 6) assess severity of pain and 7 items (questions 9A to 9G) assess interference of pain. The pain interference subscale score was determined by calculating the mean of responses to Q9A - Q9G [Q9A (general activity), Q9B (mood),Q9C (walking), Q9D (working), Q9E (relations with others), Q9F (sleep), and Q9G (enjoyment of life)] and the severity of pain subscale score was determined by calculating the mean of responses to Q3 - Q6 [Q3 (worst pain in last 24 hours), Q4 (least pain in last 24 hours), Q5 (average pain), and Q6 ("pain right now")]. A lower score indicates lower pain.
Time Frame: Up to 52 weeks in the Core Study maintenance period, and up to 24 weeks in the Extension Period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 721 | 106
units on a scale
  General Activity (Q9A) | 3.24 (2.205) | 3.27 (2.063)
  Mood (Q9B) | 2.23 (2.094) | 1.90 (1.825)
  Walking Ability (Q9C) | 3.07 (2.402) | 2.98 (2.298)
  Normal Work (Q9D) | 3.22 (2.346) | 3.21 (2.212)
  Relations with Others (Q9E) | 1.63 (1.934) | 1.34 (1.620)
  Sleep (Q9F) | 2.63 (2.258) | 2.43 (1.931)
  Enjoyment of Life (Q9G) | 2.55 (2.312) | 2.23 (2.086)
  BPI - Pain Interference Subscale Score | 2.65 (2.011) | 2.48 (1.783)
  Worst Pain - Last 24 Hours (Q3) | 4.52 (1.966) | 4.71 (1.875)
  Least Pain - Last 24 Hours (Q4) | 2.88 (1.741) | 2.90 (1.494)
  Average Pain (Q5) | 3.67 (1.703) | 3.72 (1.560)
  Pain Right Now (Q6) | 3.39 (1.846) | 3.49 (1.606)
  BPI - Severity of Pain Subscale Score | 3.62 (1.730) | 3.71 (1.562)

6. Secondary Outcome: Medical Outcomes Study 36-item Short Form (SF-36)
Description: The SF-36 is a generic health survey with 36 items that measure functional health and well-being from the subject's perspective. The 36 questions are grouped into 11 sections. Some of the sections consist of multiple questions. The survey is summarized into 8 dimensions/scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. From the 8 health dimensions, physical component summary, and mental component summary measures are derived. Scores on each scale ranged from 0 to 100; a higher score indicates a better perception of health.
Time Frame: Up to 52 weeks in the Core Study maintenance period, and up to 24 weeks in the Extension Period
Population: The Core Study population analyzed was the group of subjects who received at least 1 dose of study drug during the maintenance period and provided data. The Extension Period safety population was the group of core study safety population subjects who entered the extension period and received at least 1 dose of study drug in the extension period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 717 | 106
units on a scale
  Physical Functioning | 40.61 (9.709) | 41.93 (9.258)
  Role Physical | 43.27 (8.585) | 43.78 (8.545)
  Bodily Pain | 42.54 (6.859) | 43.05 (6.608)
  General Health | 49.28 (9.979) | 49.18 (10.498)
  Vitality | 49.77 (9.473) | 50.45 (9.109)
  Social Functioning | 49.44 (7.992) | 50.55 (7.055)
  Role Emotional | 50.63 (7.570) | 51.60 (7.109)
  Mental Health | 52.75 (8.060) | 52.93 (8.199)
  Physical Component Summary | 40.38 (8.962) | 41.04 (8.809)
  Mental Component Summary | 55.13 (8.638) | 55.68 (8.506)

7. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC is an ordinal scale of global evaluation that assesses the change in overall status relative to the start of the study. The scale has only 1 item that measures global change of overall status (improvement or worsening) by the subject on a 7-point scale (Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse.
Time Frame: At Week 52 in the Core Study maintenance period and at Week 24 in the Extension Period
Population: The Core Study population analyzed was the group of subjects who received at least 1 dose of study drug during the study. The Extension Period safety population was the group of core study safety population subjects who entered the extension period and received at least 1 dose of study drug in the extension period.
Measure: Number; unit: participants
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 773 | 105
participants
  Very much improved | 132 | 21
  Much improved | 276 | 55
  Minimally improved | 164 | 17
  No change | 121 | 9
  Minimally worse | 47 | 2
  Much worse | 29 | 1
  Very much worse | 4 | 0

8. Secondary Outcome: Treatment Satisfaction Questionnaire (TSQ) - Part I
Description: The TSQ is a self-administered questionnaire that consists of 2 parts. Part I has 6 questions (Q1 to Q6) that ask the subject to rate the experience with use of the study drug in comparison to the prestudy pain medication regarding ease of use, convenience, frequency, pain control, and overall satisfaction. Each question was rated on a scale from 1 (extremely satisfied) to 6 (extremely dissatisfied): Q1=Satisfaction with study drug; Q2=Ease of study drug use to treat pain; Q3=Convenience of study drug to treat pain; Q4=Overall drug satisfaction managing pain; Q5=Satisfaction with frequency of use; Q6=Ease of planning study drug use. The number of subjects with each category (1-6) of response for each individual question (Q1-Q6) was summarized for subjects who entered the core study maintenance period and responded to each question. TSQ - Part I was not administered in the extension period.
Time Frame: At Week 52 or upon early discontinuation at or before Week 4 in the Core Study maintenance period
Population: The Core Study population analyzed was the group of subjects who received at least 1 dose of study drug during the maintenance period and provided data.
Measure: Number; unit: participants
Arm/Group | HYD Core Study
Number analyzed (Participants) | 728
participants
  Q1: Satisfaction - extremely satisfied: number analyzed (Participants) | 593
  Q1: Satisfaction - extremely satisfied | 140
  Q1: very satisfied: number analyzed (Participants) | 593
  Q1: very satisfied | 220
  Q1: satisfied: number analyzed (Participants) | 593
  Q1: satisfied | 181
  Q1: dissatisfied: number analyzed (Participants) | 593
  Q1: dissatisfied | 38
  Q1: very dissatisfied: number analyzed (Participants) | 593
  Q1: very dissatisfied | 8
  Q1: extremely dissatisfied: number analyzed (Participants) | 593
  Q1: extremely dissatisfied | 6
  Q2: Ease of study drug use - extremely easy: number analyzed (Participants) | 593
  Q2: Ease of study drug use - extremely easy | 253
  Q2: very easy: number analyzed (Participants) | 593
  Q2: very easy | 209
  Q2: easy: number analyzed (Participants) | 593
  Q2: easy | 110
  Q2: difficult: number analyzed (Participants) | 593
  Q2: difficult | 15
  Q2: very difficult: number analyzed (Participants) | 593
  Q2: very difficult | 4
  Q2: extremely difficult: number analyzed (Participants) | 593
  Q2: extremely difficult | 2
  Q3: Convenience of study drug-extremely convenient: number analyzed (Participants) | 593
  Q3: Convenience of study drug-extremely convenient | 266
  Q3: very convenient: number analyzed (Participants) | 593
  Q3: very convenient | 196
  Q3: convenient: number analyzed (Participants) | 593
  Q3: convenient | 118
  Q3: inconvenient: number analyzed (Participants) | 593
  Q3: inconvenient | 8
  Q3: very inconvenient: number analyzed (Participants) | 593
  Q3: very inconvenient | 4
  Q3: extremely inconvenient: number analyzed (Participants) | 593
  Q3: extremely inconvenient | 1
  Q4: Overall drug satisfaction- extremely satisfied: number analyzed (Participants) | 593
  Q4: Overall drug satisfaction- extremely satisfied | 141
  Q4: very satisfied: number analyzed (Participants) | 593
  Q4: very satisfied | 200
  Q4: satisfied: number analyzed (Participants) | 593
  Q4: satisfied | 195
  Q4: dissatisfied: number analyzed (Participants) | 593
  Q4: dissatisfied | 44
  Q4: very dissatisfied: number analyzed (Participants) | 593
  Q4: very dissatisfied | 6
  Q4: extremely dissatisfied: number analyzed (Participants) | 593
  Q4: extremely dissatisfied | 7
  Q5: Satisfaction use frequency-extremely satisfied: number analyzed (Participants) | 593
  Q5: Satisfaction use frequency-extremely satisfied | 265
  Q5: very satisfied: number analyzed (Participants) | 593
  Q5: very satisfied | 169
  Q5: satisfied: number analyzed (Participants) | 593
  Q5: satisfied | 139
  Q5: dissatisfied: number analyzed (Participants) | 593
  Q5: dissatisfied | 14
  Q5: very dissatisfied: number analyzed (Participants) | 593
  Q5: very dissatisfied | 4
  Q5: extremely dissatisfied: number analyzed (Participants) | 593
  Q5: extremely dissatisfied | 2
  Q6: Ease of planning use - extremely easy: number analyzed (Participants) | 593
  Q6: Ease of planning use - extremely easy | 284
  Q6: very easy: number analyzed (Participants) | 593
  Q6: very easy | 189
  Q6: easy: number analyzed (Participants) | 593
  Q6: easy | 106
  Q6: difficult: number analyzed (Participants) | 593
  Q6: difficult | 11
  Q6: very difficult: number analyzed (Participants) | 593
  Q6: very difficult | 1
  Q6: extremely difficult: number analyzed (Participants) | 593
  Q6: extremely difficult | 2

9. Secondary Outcome: Treatment Satisfaction Questionnaire (TSQ) - Part II
Description: The TSQ is a self-administered questionnaire that consists of 2 parts. Part II has 2 questions that measure the subject's willingness to continue the use of study drug as pain medication (Q1), and to recommend the study drug to someone else (Q2). Question 1 consists of 6 categories of response rated on a scale from 1 (very willing to continue) to 6 (very unwilling to continue): 1=Very willing to continue; 2=Willing to continue; 3=Somewhat willing to continue; 4=Somewhat unwilling to continue; 5=Unwilling to continue; 6=Very unwilling to continue. Question 2 consists of 3 categories of response: 1=yes; 2=no; 3=undecided. The number of subjects with each category of response for each individual question was summarized for subjects completing the core study maintenance period and for those enrolled in the extension period.
Time Frame: At Week 52 or upon early discontinuation at or before Week 4 in maintenance and at Week 24 in extension
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | HYD Core Study | HYD Extension Period
Number analyzed (Participants) | 728 | 106
participants
  Q1:Willingness to continue study drug-very willing: number analyzed (Participants) | 636 | 105
  Q1:Willingness to continue study drug-very willing | 281 | 51
  Q1: willing to continue: number analyzed (Participants) | 636 | 105
  Q1: willing to continue | 141 | 29
  Q1: somewhat willing to continue: number analyzed (Participants) | 636 | 105
  Q1: somewhat willing to continue | 53 | 18
  Q1: somewhat unwilling to continue: number analyzed (Participants) | 636 | 105
  Q1: somewhat unwilling to continue | 29 | 4
  Q1: unwilling to continue: number analyzed (Participants) | 636 | 105
  Q1: unwilling to continue | 79 | 3
  Q1: very unwilling to continue: number analyzed (Participants) | 636 | 105
  Q1: very unwilling to continue | 53 | 0
  Q2: Recommend study drug for pain - yes: number analyzed (Participants) | 636 | 105
  Q2: Recommend study drug for pain - yes | 546 | 90
  Q2: no: number analyzed (Participants) | 636 | 105
  Q2: no | 36 | 4
  Q2: undecided: number analyzed (Participants) | 636 | 105
  Q2: undecided | 54 | 11

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from start of study participation through the period beyond study completion: up to 84 weeks.
Description: AEs were learned of through spontaneous reports and/or subject interview, or observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or 30 days after last study drug dose. Serious AEs up to 30 days after last study drug dose or last visit were followed until AE or sequelae resolved/stabilized.
Arm/Group | HYD Core Study | HYD Extension Period
Serious Adverse Events (participants affected / at risk) | 80/922 | 6/106
Other Adverse Events (participants affected / at risk) | 586/922 | 0/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HYD Core Study (N=922) | HYD Extension Period (N=106)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 — Outcome: Death. 1 subject experienced 2 serious AEs resulting in death: thrombotic thrombocytopenic purpura and metabolic acidosis.
Acute myocardial infarction (Cardiac disorders) | 1 | 0 — Outcome: Death
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 5 | 1
Device dislocation (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 — Outcome: Death
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 — Outcome: Death 1 subject experienced 2 serious AEs resulting in death: thrombotic thrombocytopenic purpura and metabolic acidosis.
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleomorphic liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 5 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Outcome: Death
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Outcome: Death
Abortion induced (Surgical and medical procedures) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HYD Core Study (N=922) | HYD Extension Period (N=106)
Nausea (Gastrointestinal disorders) | 218 | 0
Constipation (Gastrointestinal disorders) | 193 | 0
Vomiting (Gastrointestinal disorders) | 100 | 0
Diarrhoea (Gastrointestinal disorders) | 56 | 0
Fatigue (General disorders) | 71 | 0
Upper respiratory tract infection (Infections and infestations) | 73 | 0
Sinusitis (Infections and infestations) | 50 | 0
Nasopharyngitis (Infections and infestations) | 47 | 0
Urinary tract infection (Infections and infestations) | 47 | 0
Dizziness (Nervous system disorders) | 106 | 0
Somnolence (Nervous system disorders) | 104 | 0
Headache (Nervous system disorders) | 85 | 0
Insomnia (Psychiatric disorders) | 57 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 52 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days